CLINICAL TRIAL: NCT04363021
Title: Is a History of Pre-eclampsia Before Systemic Sclerosis Onset a Risk Factor for Vascular Phenotype in Women With Systemic Sclerosis?
Brief Title: Is a History of Pre-eclampsia a Risk Factor for Vascular Phenotype in Women With Systemic Sclerosis?
Acronym: PREVASCLERO
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PREVASCLERO (29BRC20.0080)
Record Dates: First submitted 2020-04-20; First posted 2020-04-27 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Systemic Sclerosis; Preeclampsia; Vascular Complications
Keywords: systemic sclerosis; vascular phenotype; pre-eclampsia
MeSH Terms: conditions — Scleroderma, Systemic; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: Cases will be defined as women with systemic sclerosis, specific vascular complications (digital ulcers, specific cardiac involvement of systemic sclerosis including pulmonary arterial hypertension, renal crisis) and with a previous pregnancy longer than 6 months before systemic sclerosis diagnosis.
- controls: Controls will be defined as women with systemic sclerosis, no specific vascular complication and with a previous pregnancy longer than 6 months before systemic sclerosis diagnosis.

SUMMARY:
Background:

Pre-eclampsia, defined by the association of an arterial hypertension and significant proteinuria after 20 weeks of gestation, complicates 1 to 2% of pregnancies in France. Its pathophysiology involves angiogenesis impairment, upregulated maternal systemic inflammatory response, activation of oxidative stress and endothelial dysfunction.

In a recent Danish nation-wide cohort study, pre-eclampsia was associated with a 69% increased risk of later developing scleroderma.

Type of study: prospective observational case-control study. Primary objective of the study: to determine if a history of pre-eclampsia before systemic sclerosis diagnosis is an independent risk factor for vascular phenotype in sclerodermic women.

Secondary objective: to describe all risk factors for vascular phenotype in sclerodermic women with a previous pregnancy longer than 6 months before scleroderma diagnosis.

DETAILED DESCRIPTION:
Background :

Pre-eclampsia is defined by the association of an arterial hypertension and significant proteinuria after 20 weeks of gestation. It complicates 1 to 2% of pregnancies in France. Its pathophysiology involves angiogenesis impairment, upregulated maternal systemic inflammatory response, activation of oxidative stress and endothelial dysfunction.

In a recent Danish nation-wide cohort study, pre-eclampsia was associated with a 69% increased risk of later developing scleroderma. A case-control study on 103 women with systemic sclerosis compared to 103 control women had already found an increased incidence of previous vasculoplacental disorders in women with systemic sclerosis. Women developed systemic sclerosis on average 27 years after their first pregnancy.

Primary objective of the study : to determine if a history of pre-eclampsia before systemic sclerosis diagnosis is an independent risk factor for vascular phenotype in sclerodermic women.

Secondary objective: to describe all risk factors for vascular phenotype in sclerodermic women with a previous pregnancy longer than 6 months before scleroderma diagnosis.

Conduct of the study:

It is a prospective observational case-control study. Cases will be defined as women with systemic sclerosis, specific vascular complications (digital ulcers, specific cardiac involvement of systemic sclerosis including pulmonary arterial hypertension, renal crisis) and with a previous pregnancy longer than 6 months before systemic sclerosis diagnosis.

Controls will be defined as women with systemic sclerosis, no specific vascular complication and with a previous pregnancy longer than 6 months before systemic sclerosis diagnosis.

Conduct of the study:

A self-administered " pregnancy " questionnaire will be given to each women with systemic sclerosis of the cohort group during the annual follow-up consultation. A case report form will be completed at the same time by the physician in charge of the patient.

The " pregnancy " questionnaire will consist of two parts :

* A part " pre-eclampsia questionnaire ", derived from the translation in French of a questionnaire validated in English.
* A second part with additional questions on pregnancies. The duration of participation to the study will be of one day. The duration of the inclusion period will be of 24 months. Needed number of patients : 378 women, 126 "cases" and 252 "control" .

Perspectives of the study :

If this study demonstrates that a previous pre-eclampsia is an independent risk factor for vascular phenotype in women with systemic sclerosis, it will be mandatory to look for a history of pre-eclampsia in women at the time of systemic sclerosis diagnosis. Besides, the women with a history of pre-eclampsia should be monitored more frequently for vascular complications related to systemic sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* General:

Women with a diagnosis of systemic sclerosis according to EULAR 2013 diagnostic criteria AND with a history of pregnancy longer than 6 months (28 weeks of gestation (WG)) before systemic sclerosis diagnosis.

* Specific:

For the women of the " case " group :

Women with vascular complications specific of systemic sclerosis (digital ulcers, specific cardiac involvement of systemic sclerosis including pulmonary arterial hypertension, renal crisis).

For the women of the " control " group :

Women with no vascular complications specific of systemic sclerosis.

Non inclusion criteria :

* Refusal to participate to the study
* Minor women
* Women under tutorship
* Women with no pregnancy history or with a history of pregnancy(ies) below 6 months length.

Exclusion Criteria:

* Women aged of less than 18 years
* Women on legal protection
* Women with no history of pregnancy of more than 6 months
* Women unable to fill out a questionnaire in French
* Women who refuse to participate to the study

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women with a diagnosis of systemic sclerosis according to EULAR 2013 diagnostic criteria AND with a history of pregnancy longer than 6 months (28 WG) before systemic sclerosis diagnosis
  followed in one of the French centers of expertise for systemic sclerosis will be offered to participate to the study during the annual follow-up consultation with her referring physician.
Sampling Method: Non-Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
History of pre-eclampsia before systemic sclerosis diagnosis | Inclusion (Day 0)
  Primary outcome will be evaluated by the proportion of women with a history of pre-eclampsia before systemic sclerosis diagnosis in each group. Primary judgement criterion will be the response of a woman to the " pre-eclampsia questionnaire ". The aim is to determine if a history of pre-eclampsia before systemic sclerosis diagnosis is an independent prognostic factor for vascular phenotype in sclerodermic women.
  Primary judgement criterion: Responses of the women to the " pre-eclampsia questionnaire ".

SECONDARY OUTCOMES:
Risk factors for vascular phenotype in sclerodermic women with a previous pregnancy longer than 6 months | Inclusion (Day 0)
  Secondary outcomes will be evaluated by the proportion of women with chronic hypertension, diffuse systemic sclerosis, disease duration > 5 years, anti-centromere antibodies, anti-Scl70 antibodies, antiphospholipid antibodies, antiphospholipid syndrome, interstitial lung disease, and tobacco use, in each group, mean age at systemic sclerosis diagnosis in each group. Secondary judgement criteria will be patients' clinical, biological and radiological medical data. The aim is to describe all risk factors for vascular phenotype in sclerodermic women with a previous pregnancy longer than 6 months.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Dijon, Dijon
  - CHU de Lille, Lille
  - CHU de Limoges, Limoges
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - CHU de Rennes, Rennes
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning two year and ending five years following the end study
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Background] Societe francaise d'anesthesie et de reanimation (Sfar); College national des gynecologues et obstetriciens francais (CNGOF); Societe francaise de medecine perinatale (SFMP); Societe francaise de neonatalogie (SFNN). [Multidisciplinary management of severe pre-eclampsia (PE). Experts' guidelines 2008. Societe francaise d'anesthesie et de reanimation. College national des gynecologues et obstetriciens francais. Societe francaise de medecine perinatale. Societe francaise de neonatalogie]. Ann Fr Anesth Reanim. 2009 Mar;28(3):275-81. doi: 10.1016/j.annfar.2009.02.015. Epub 2009 Mar 24. No abstract available. French. PMID 19321292
- [Background] Saucedo M, Deneux-Tharaux C, Bouvier-Colle MH; Le Comite national d'experts sur la mortalite maternelle. [Maternal mortality in France, 2007-2009]. J Gynecol Obstet Biol Reprod (Paris). 2013 Nov;42(7):613-27. doi: 10.1016/j.jgyn.2013.06.011. Epub 2013 Sep 13. French. PMID 24035736
- [Background] Conrad KP, Miles TM, Benyo DF. Circulating levels of immunoreactive cytokines in women with preeclampsia. Am J Reprod Immunol. 1998 Aug;40(2):102-11. doi: 10.1111/j.1600-0897.1998.tb00398.x. PMID 9764352
- [Background] Redman CW, Sargent IL. Pre-eclampsia, the placenta and the maternal systemic inflammatory response--a review. Placenta. 2003 Apr;24 Suppl A:S21-7. doi: 10.1053/plac.2002.0930. PMID 12842410
- [Background] Zhou CC, Zhang Y, Irani RA, Zhang H, Mi T, Popek EJ, Hicks MJ, Ramin SM, Kellems RE, Xia Y. Angiotensin receptor agonistic autoantibodies induce pre-eclampsia in pregnant mice. Nat Med. 2008 Aug;14(8):855-62. doi: 10.1038/nm.1856. Epub 2008 Jul 27. PMID 18660815
- [Background] Herse F, Verlohren S, Wenzel K, Pape J, Muller DN, Modrow S, Wallukat G, Luft FC, Redman CW, Dechend R. Prevalence of agonistic autoantibodies against the angiotensin II type 1 receptor and soluble fms-like tyrosine kinase 1 in a gestational age-matched case study. Hypertension. 2009 Feb;53(2):393-8. doi: 10.1161/HYPERTENSIONAHA.108.124115. Epub 2008 Dec 8. PMID 19064815
- [Background] Lim R, Acharya R, Delpachitra P, Hobson S, Sobey CG, Drummond GR, Wallace EM. Activin and NADPH-oxidase in preeclampsia: insights from in vitro and murine studies. Am J Obstet Gynecol. 2015 Jan;212(1):86.e1-12. doi: 10.1016/j.ajog.2014.07.021. Epub 2014 Jul 18. PMID 25046804
- [Background] Roberts JM, Taylor RN, Musci TJ, Rodgers GM, Hubel CA, McLaughlin MK. Preeclampsia: an endothelial cell disorder. Am J Obstet Gynecol. 1989 Nov;161(5):1200-4. doi: 10.1016/0002-9378(89)90665-0. PMID 2589440
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams DJ. Pre-eclampsia and risk of cardiovascular disease and cancer in later life: systematic review and meta-analysis. BMJ. 2007 Nov 10;335(7627):974. doi: 10.1136/bmj.39335.385301.BE. Epub 2007 Nov 1. PMID 17975258
- [Background] Kamper-Jorgensen M, Gammill HS, Nelson JL. Preeclampsia and scleroderma: a prospective nationwide analysis. Acta Obstet Gynecol Scand. 2018 May;97(5):587-590. doi: 10.1111/aogs.13296. Epub 2018 Feb 8. PMID 29344946
- [Background] van Wyk L, van der Marel J, Schuerwegh AJ, Schouffoer AA, Voskuyl AE, Huizinga TW, Bianchi DW, Scherjon SA. Increased incidence of pregnancy complications in women who later develop scleroderma: a case control study. Arthritis Res Ther. 2011;13(6):R183. doi: 10.1186/ar3510. Epub 2011 Nov 4. PMID 22053948
- [Background] Englert H, Small-McMahon J, Davis K, O'Connor H, Chambers P, Brooks P. Systemic sclerosis prevalence and mortality in Sydney 1974-88. Aust N Z J Med. 1999 Feb;29(1):42-50. doi: 10.1111/j.1445-5994.1999.tb01587.x. PMID 10200812
- [Background] Lee P, Langevitz P, Alderdice CA, Aubrey M, Baer PA, Baron M, Buskila D, Dutz JP, Khostanteen I, Piper S, et al. Mortality in systemic sclerosis (scleroderma). Q J Med. 1992 Feb;82(298):139-48. PMID 1620814
- [Background] Simeon CP, Armadans L, Fonollosa V, Solans R, Selva A, Villar M, Lima J, Vaque J, Vilardell M. Mortality and prognostic factors in Spanish patients with systemic sclerosis. Rheumatology (Oxford). 2003 Jan;42(1):71-5. doi: 10.1093/rheumatology/keg033. PMID 12509616
- [Background] Jacobsen S, Halberg P, Ullman S. Mortality and causes of death of 344 Danish patients with systemic sclerosis (scleroderma). Br J Rheumatol. 1998 Jul;37(7):750-5. doi: 10.1093/rheumatology/37.7.750. PMID 9714351
- [Background] Hesselstrand R, Scheja A, Akesson A. Mortality and causes of death in a Swedish series of systemic sclerosis patients. Ann Rheum Dis. 1998 Nov;57(11):682-6. doi: 10.1136/ard.57.11.682. PMID 9924211
- [Background] LeRoy EC, Black C, Fleischmajer R, Jablonska S, Krieg T, Medsger TA Jr, Rowell N, Wollheim F. Scleroderma (systemic sclerosis): classification, subsets and pathogenesis. J Rheumatol. 1988 Feb;15(2):202-5. No abstract available. PMID 3361530
- [Background] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Csuka ME, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American College of Rheumatology/European League against Rheumatism collaborative initiative. Arthritis Rheum. 2013 Nov;65(11):2737-47. doi: 10.1002/art.38098. Epub 2013 Oct 3. PMID 24122180
- [Background] Riemekasten G, Philippe A, Nather M, Slowinski T, Muller DN, Heidecke H, Matucci-Cerinic M, Czirjak L, Lukitsch I, Becker M, Kill A, van Laar JM, Catar R, Luft FC, Burmester GR, Hegner B, Dragun D. Involvement of functional autoantibodies against vascular receptors in systemic sclerosis. Ann Rheum Dis. 2011 Mar;70(3):530-6. doi: 10.1136/ard.2010.135772. Epub 2010 Nov 15. PMID 21081526
- [Background] Walther T, Wallukat G, Jank A, Bartel S, Schultheiss HP, Faber R, Stepan H. Angiotensin II type 1 receptor agonistic antibodies reflect fundamental alterations in the uteroplacental vasculature. Hypertension. 2005 Dec;46(6):1275-9. doi: 10.1161/01.HYP.0000190040.66563.04. Epub 2005 Oct 31. PMID 16260641
- [Background] Nelson JL, Furst DE, Maloney S, Gooley T, Evans PC, Smith A, Bean MA, Ober C, Bianchi DW. Microchimerism and HLA-compatible relationships of pregnancy in scleroderma. Lancet. 1998 Feb 21;351(9102):559-62. doi: 10.1016/S0140-6736(97)08357-8. PMID 9492775
- [Background] Allanore Y, Distler O, Matucci-Cerinic M, Denton CP. Review: Defining a Unified Vascular Phenotype in Systemic Sclerosis. Arthritis Rheumatol. 2018 Feb;70(2):162-170. doi: 10.1002/art.40377. Epub 2018 Jan 22. PMID 29145709
- [Background] Lescoat A, Yelnik CM, Coiffier G, Wargny M, Lamotte C, Cazalets C, Belhomme N, Ballerie A, Hatron PY, Launay D, Perdriger A, Sobanski V, Hachulla E, Jego P. Ulnar Artery Occlusion and Severity Markers of Vasculopathy in Systemic Sclerosis: A Multicenter Cross-Sectional Study. Arthritis Rheumatol. 2019 Jun;71(6):983-990. doi: 10.1002/art.40799. Epub 2019 Apr 29. PMID 30552835
- [Background] Diehl CL, Brost BC, Hogan MC, Elesber AA, Offord KP, Turner ST, Garovic VD. Preeclampsia as a risk factor for cardiovascular disease later in life: validation of a preeclampsia questionnaire. Am J Obstet Gynecol. 2008 May;198(5):e11-3. doi: 10.1016/j.ajog.2007.09.038. Epub 2008 Feb 1. PMID 18241822